CLINICAL TRIAL: NCT00356720
Title: Clinical Efficacy and Safety of 2 Dosing Regimens of T1225 Eye Drops 1.5% (Instilled Twice Daily for 2 or 3 Days) Versus Oral Azithromycin in Treatment of Trachoma
Brief Title: Efficacy and Safety of 2 Dosing Regimens of T1225 Eye Drops 1.5% Versus Oral Azithromycin in Treatment of Trachoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT1225-PIII-10/03
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2006-07-26 (Estimated); Status verified 2006-07

CONDITIONS: Trachoma
MeSH Terms: conditions — Trachoma | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To assess in children the efficacy and safety of 2 dosing regimens of T1225 1.5% eye drops, in comparison to a reference product, single-dose oral azithromycin (AZM) 20 mg/kg, for the treatment of active trachoma. Evaluation of clinical efficacy was primary (% of clinical cure at Day 60 in Per Protocol Set), microbiological evaluation was secondary

DETAILED DESCRIPTION:
The aim of the present study was to compare the efficacy of the dosing regimen which was demonstrated in pharmacokinetic studies to be the best candidate for trachoma treatment (T1225 1.5% eye drops BID for 3 days) with a shorter duration of treatment (T1225 1.5% eye drops BID for 2 days) and with a single oral administration of AZM (20 mg/kg) in patients suffering from active trachoma. The study was to be performed in approximately 600 children (aged 1 to 10 years) from Guinea Conakry and Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 1-10 years;
* written informed consent by legally acceptable representative;
* TF+ TI0 (trachomatous inflammation - follicular) or TF+TI+ (trachomatous inflammation - follicular and intense) on simplified World Health Organisation (WHO) grading system

Exclusion Criteria:

* Trichiasis or corneal opacity;
* palpebral deformation;
* clinically significant ocular abnormality;
* ocular infection;
* organic amblyopia;
* hypersensitivity to treatments' components;
* immunosuppressive conditions;
* systemic AZM or steroids;
* topical ophthalmic antibiotics within 3 months;
* other systemic antibiotics within 1 month;
* topical (ocular, nasal, bronchial etc.) treatments within 1 week;
* systemic non-steroidal anti-inflammatory drugs on day before Day 0

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2004-01; Study Completion 2004-05

PRIMARY OUTCOMES:
Cure at end of study, i.e. TF0 grade on simplified WHO trachoma grading system < 5 follicles ≥ 0.5 mm diameter in upper tarsal conjunctiva) in the worse eye
at the end of the study

SECONDARY OUTCOMES:
Cure at Days 30 and 60,
cure in both eyes,
trachoma grades at each visit;
microbiological cure;
Ocular signs (bulbar conjunctival hyperaemia, discharge; lachrymation;
Global efficacy assessment by investigator.
Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle COCHEREAU, Professor, Principal Investigator — CHU d'Angers, France